CLINICAL TRIAL: NCT03007303
Title: The Relevance Between the microRNA-30e in Plasma and the Prognosis of Schizophrenia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dalian Seventh People's Hospital (Other)
Collaborators: TAKARA BIOTECHNOLOGY(DALIAN)CO.,LTD. (Unknown)
Responsible Party: Principal Investigator, Shoufu Xie, chief physician，Professor of Psychiatry,Vice president of the hospital, Dalian Seventh People's Hospital
Other Study IDs: GFu01
Record Dates: First submitted 2016-11-17; First posted 2017-01-02 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia; Micrognathia
MeSH Terms: conditions — Schizophrenia; Micrognathism | interventions — Olanzapine; Quetiapine Fumarate; ziprasidone; Risperidone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Biospecimen Retention: Samples With DNA — The peripheral blood sample Plasma separated from the peripheral blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- schizophrenia: 15 patients with schizophrenia will be treated with anyone of the atypical psychotics(including olanzapine, quetiapine , ziprasidone and risperidone)or combined with MECT.
  The fluctuating dosage depends on the changes of symptom according to the total scores of Positive and Negative Syndrome Scale from schizophrenia patients after treated.
  Interventions: Drug: Atypical Antipsychotic; Other: atypical antipsychotic combined with MECT
- health controls: 15 healthy individuals were collected from Dalian seventh people's hospital and were matched on age and sex to schizophrenia group

INTERVENTIONS:
Drug: Atypical Antipsychotic — Olanzapine: tablet ,5-20mg, Po q.d. Risperidone: tablet ,1-3 mg, Po q.d. Quetiapine: tablet ,100-400mg, Po b.i.d. ziprasidone : tablet ,40 -80mg, Po b.i.d.
  Other Names: olanzapine, quetiapine , ziprasidone and risperidone
  Groups: schizophrenia
Other: atypical antipsychotic combined with MECT — The schizophrenia who matches the indications such as severe negativism, refused to eating or stupor may be treated with antipsychotic combined with MECT, the frequency and times of MECT depend on the state of illness
  Other Names: MECT means modified electric convulsive therapy
  Groups: schizophrenia

SUMMARY:
This study investigates the relationship of circulating microRNA-30e and schizophrenia, and shows the relevance of the aberrant microRNA-30e expression in plasma with the variation disease status.

DETAILED DESCRIPTION:
The plasma samples from 15 individuals with schizophrenia (with a diagnosis of ICD-10) and the equivalent healthy controls will be conducted with the quantification analysis of the microRNA-30e via real-time quantitative polymerase chain reaction(RT-PCR).

The 15 patients enrolled should be the first-episode and have not been treated, or were drug free 3 months recently at least.

This research measures the expression level of microRNA-30e in schizophrenia respectively before the beginning treatment with atypical psychotics or combined with MECT, after the 4-week treated , the 8-week treated compared with 15 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Persons should be diagnosed with schizophrenia according to the International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10)
* The first-onset or drug-free in the latest 3 months
* Between the ages of 17-40

Exclusion Criteria:

* Comorbid with other psychosis
* Have physical or neurological diseases such as traumatic brain injuries
* History of drug-abused or alcoholic
* Blood transfusion history in a month
* Been treated with Modified Electric Convulsive Therapy(MECT) in late 3 months

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: the first-onset schizophrenia patients or drug-free suffers in the last 3 months，who are Chinese of Han descent and admitted to the Dalian Seventh People's Hospital,China
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-03 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
the Baseline expression profiling of microRNA-30e measured by real-time quantitative poly-chain reaction (QPCR) | before the treatment
  the plasma samples will be collected from the patients with schizophrenia and the healthy controls at the beginning recruit for the microRNA-30e detection
the Changed expression level of microRNA-30e measured by real-time quantitative poly-chain reaction (QPCR) | Change from Baseline expression level at 4-week treatment
  the plasma samples will be collected from the patients with schizophrenia at the 4-week treatment for the microRNA-30e detection
the Changed expression level of microRNA-30e measured by real-time quantitative poly-chain reaction (QPCR) | Change from Baseline expression level at 8-week treatment
  the plasma samples will be collected from the patients with schizophrenia at the 8-week treatment for the microRNA-30e detection

SECONDARY OUTCOMES:
the scores of Positive and Negative Syndrome Scale(PANSS) for the patients with schizophrenia | before, after 4 weeks and 8 weeks treatment
  The PANSS for estimating the severity of positive and negative symptoms in schizophrenia
The degree of Personal and Social Performance scale(PSP) for the patients with schizophrenia | before, after 4 weeks and 8 weeks treatment
  The degree of Personal and Social Performance scale(PSP) used to evaluate the disable levels in Multiple dimensions ,especially in social and self-care performance
The scale of Clinical Global Impression(CGI) in patients with schizophrenia after treatment | 4 weeks and 8 weeks treatment
  Main purpose to provide a global rating of illness severity ,improvement and response to treatment for the patients with schizophrenia

CONTACTS AND LOCATIONS:
Overall Officials: Shoufu Xie, postgraduate, Principal Investigator — Dalian Seventh People's Hospital
Locations (1):
- Dalian Seventh People's Hospital, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Xu C, Liu X, Song X, Gao Q, Cheng L, Wang L, Zhang K, Xu Y. Aberrant resting state in microRNA-30e rat model of cognitive impairment. Neuroreport. 2016 Aug 3;27(11):809-17. doi: 10.1097/WNR.0000000000000616. PMID 27258654
- [Result] Xu Y, Li F, Zhang B, Zhang K, Zhang F, Huang X, Sun N, Ren Y, Sui M, Liu P. MicroRNAs and target site screening reveals a pre-microRNA-30e variant associated with schizophrenia. Schizophr Res. 2010 Jun;119(1-3):219-27. doi: 10.1016/j.schres.2010.02.1070. Epub 2010 Mar 27. PMID 20347265
- [Result] Banigan MG, Kao PF, Kozubek JA, Winslow AR, Medina J, Costa J, Schmitt A, Schneider A, Cabral H, Cagsal-Getkin O, Vanderburg CR, Delalle I. Differential expression of exosomal microRNAs in prefrontal cortices of schizophrenia and bipolar disorder patients. PLoS One. 2013;8(1):e48814. doi: 10.1371/journal.pone.0048814. Epub 2013 Jan 30. PMID 23382797